CLINICAL TRIAL: NCT07022535
Title: Personalised Timing of Interval Debulking Surgery Based on KELIM After Neoadjuvant Chemotherapy in Advanced Ovarian Cancer - a Pilot Study
Brief Title: Personalised Timing of Interval Debulking Surgery in Advanced Ovarian Cancer
Acronym: PRESELECT-0
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ka-Yu Tse, Prof., The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 24-304; HKUCTR-3091 (Registry Identifier: HKU Clinical Trials Registry)
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: advanced; ovarian cancer; neoadjuvant chemotherapy; interval debulking surgery; KELIM; CA 125
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Carboplatin; Paclitaxel; Cytoreduction Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Pilot study, single-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalised management (Experimental): Patients will be managed based on CA-125 ELIMination Rate Constant K (KELIM) at the neoadjuvant setting.
  Interventions: Diagnostic Test: KELIM; Drug: Carboplatin plus Paclitaxel; Procedure: Interval debulking surgery

INTERVENTIONS:
Diagnostic Test: KELIM — (i) Patients with KELIM >=1 will receive radiological assessment and undergo interval debulking surgery if the disease is operable.
  (ii) Patients with KELIM <1 will have alternative management, such as addition of bevacizumab or changing to dose-dense chemotherapy, and defer the interval debulking surgery
Drug: Carboplatin plus Paclitaxel — Chemotherapy as neaodjuvant chemotherapy
Procedure: Interval debulking surgery — Interval debulking surgery
  Other Names: cytoreductive surgery

SUMMARY:
About 70% of epithelial ovarian cancer patients are diagnosed at advanced stage. When primary optimal surgery is not possible, neoadjuvant chemotherapy will followed by interval debulking surgery is one treatment option. However, there is no consensus on the optimal timing of the surgery. CA125 is a well-known tumor marker in ovarian cancer. Its kinetic change has been proven to correlate with the patients' response to chemotherapy and chance of optimal resection. This study aims to utilize the kinetic change of CA125 to customize the timing of surgery for individual patients.

DETAILED DESCRIPTION:
Recruited patients will have additional CA125 at 4th (before administration of chemotherapy), and 5th week after the first cycle of chemotherapy. CA-125 ELIMination Rate Constant K (KELIM) will be determined. Patients with KELIM =>1 will receive radiological assessment and undergo internal debulking surgery if the disease is operable. Patients with KELIM <1 will have alternative management, such as addition of bevacizumab or changing to dose-dense chemotherapy, and defer the interval debulking surgery

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years old.
2. Patients who have Eastern Cooperative Oncology Group (ECOG) score 0-1.
3. Patients who are competent to give informed consent.
4. Patients who have stage III-IV histologically or cytologically confirmed epithelial ovarian cancer, fallopian tube or primary peritoneal cancer not amenable for primary debulking surgery (PDS).
5. Patients who are planned for neoadjuvant chemotherapy (NACT) using platinum-based chemotherapy +/- bevacizumab or biosimilar. Those who are receiving NACT before interval debulking surgery (IDS) are also eligible.
6. Patients who have an evaluable CA125 level at baseline (i.e., baseline level is at least 2x upper limit of normal).
7. Patients who have baseline computed tomography of at least abdomen and pelvis, or positron emission tomography (PET)-CT. Magnetic resonance imaging (MRI) is also acceptable but the same modality has to be used when assessing the feasibility of IDS.
8. Patients who agree to undergo IDS, where the time of IDS may differ from the usual clinical practice.
9. Patients who agree to receive adjuvant chemotherapy, if clinically indicated. The total number of chemotherapy should be at least four or above.

Exclusion Criteria:

1. Patients who have borderline malignancy, or non-epithelial ovarian cancer like germ cell or sex cord tumor, or metastatic diseases from other origins like Krukenberg's tumor
2. Patients who are eligible for PDS
3. Patients who are not fit for PDS because of medical morbidities or refusal of operation
4. Patients who have already started NACT outside the study centres, except those who have just had one cycle within 21 days and the baseline CA125 is available.
5. Patients who are pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 18 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete resection (CC0) rate | Up to 24 months
  The likelihood of CC0 in patients who undergo IDS when KELIM reaches 1 or above
Sensitivity of KELIM in predicting CC0 | Up to 24 weeks
  The sensitivity of KELIM in predicting CC0

SECONDARY OUTCOMES:
Time required to achieve KELIM >=1 | Up to 24 weeks
  The time required for KELIM to reach >=1 in EOC patients receiving NACT
Complication rates of treatment | Up to 1 year
  The complication rates of surgery based on the Clavien-Dindo classification and chemotherapy based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Quality-of-life scale | Up to 1 year
  Different functional scales will be assessed by questionnaires like the EORTC questionnaires where all scales range from 0-100. The higher the score, the greater the intensity of that particular item is.

OTHER OUTCOMES:
Expression of biomarkers | Up to 1 year
  Expression levels of biomarkers before and after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yu Tse, MBBS, MMedSc, PhD, FRCOG, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Patients' disease course based on this novel management algorithm
Supporting Information: Study Protocol
Time Frame: One year after the end of the study
Access Criteria: The study protocol will be available under a reasonable request to the corresponding author